CLINICAL TRIAL: NCT03044054
Title: Treatment of Breast Fibroadenoma Targeted Tissue With High Intensity Focused Ultrasound (HIFU)
Brief Title: Treatment of Breast Fibroadenoma Targeted Tissue With HIFU
Acronym: HIFU-003
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/FA/003
Record Dates: First submitted 2017-01-17; First posted 2017-02-06 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Fibroadenoma
Keywords: HIFU
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECHOPULSE (Experimental): ECHOPULSE HIFU
  Interventions: Device: ECHOPULSE

INTERVENTIONS:
Device: ECHOPULSE — HIFU Under ultrasound guidance

SUMMARY:
This study evaluates the efficacy and the safety of the HIFU for the treatment of breast fibroadenoma.

DETAILED DESCRIPTION:
Echopulse is specially designed, manufactured and CE marked for treating breast fibroadenoma. HIFU is a completely alternative to surgery which utilizes high-energy ultrasound to deliver a large amount of sound energy to a focal point to rapidly induce tissue heating to 85-90°C.This initiates tissue coagulation followed by tissue necrosis ablating the targeted area.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 years or older diagnosed with breast fibroadenoma and presenting at least one fibroadenoma.
2. Diagnosis of fibroadenoma must be based on:

   1. Clinical examination
   2. Ultrasound image alone for patients under 35 years old. For women older than 35 years, a mammogram will be performed in addition to ultrasound. The BI-RADS score of this mammogram must be 2 or 3. BI-RADS score of 4 is eligible if biopsy indicates fibroadenoma with concordance.
   3. Histologic confirmation by core needle biopsy.
3. Patient is a candidate for the surgery.
4. The fibroadenoma treatment volume must be at least 5 mm and no more than 26 mm from the skin. This criterion should be evaluated immediately prior treatment, once the breast is immobilized and potentially compressed.
5. The rib cage should not be in the prefocal ultrasound path or behind the target fibroadenoma (minimum distance from the posterior wall of the fibroadenoma must be at least 10 mm). This criterion shall be evaluated immediately prior to treatment, once breast is immobilized and potentially compressed.
6. The fibroadenoma is 1 cm or greater at its largest dimension and no less than 7.5 mm in the anterior-posterior dimension (measured by ultrasound). Focal point for HIFU treatment must also be at least 3 mm from any border of the fibroadenoma.
7. Patient's fibroadenoma size is greater or equal to 0.2 cc and less than 10 cc in volume (measured by ultrasound on the day of the procedure).
8. Fibroadenoma is palpable.
9. Pain ≥ 30mm/100mm measured on VAS as a maximum level during the last 30 days
10. Anxiety ≥ 30mm/100mm measured on VAS as a maximum level during the last 30 days
11. Patient has signed a written informed consent.

Exclusion Criteria:

1. Patient is pregnant or nursing.
2. Presence of calcified fibroadenoma. Calcification will be determined with mammography. In women > 35 years old, the diagnostic mammogram should be evaluated for calcification. In women ≤ 35 years old, a single view mammogram of the affected breast is sufficient for evaluation of calcification. Women ≤ 35 years old will be excluded based on the findings of calcification on a single view mammogram.
3. Patient with history of breast cancer or history of laser or radiation therapy to the target breast.
4. Patient with breast implants in the target breast.
5. Patient with a breast cyst within the fibroadenoma to be treated.
6. Patient's fibroadenoma not clearly visible on the ultrasound images (in B mode) at the inclusion visit.
7. Patient participating in another clinical trial involving an investigational drug, device or biologic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Pain level assessment | 12 Months
  visual analog scale
Anxiety level assessment | 12 Months
  visual analog scale
Volume assessment | 12 Months
  Ultrasound measurement

SECONDARY OUTCOMES:
The short (6-item) version of the State-Trait Anxiety Inventory (STAI) | inclusion visit (V0), Day 2/3, Day 7, 6 months, 12 months
Palpability of the breast fibroadenoma | inclusion visit (V0), Day 2/3, Day 7, 6 months, 12 months
  Physician clinical examination
Freedom from additional procedures for fibroadenoma of the breast | Day 2/3, Day 7, 6 months, 12 months
  Physician assessment concerning the need of additional procedures
Patient satisfaction | Month 6 and Months 12
  Self assessment satisfaction questionnaire
Safety endpoints include adverse events (AEs) and serious adverse events (SAEs) occurring at any time during the trial. | Day 0, Day 2/3, Day 7, 6 months, 12 months
  Assessment and capture of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Michel NUTA, MD, Study Director — Theraclion
Locations (4):
- United States (4):
  - Bellevue Hospital Center, New York, New York
  - New York Columbia University Medical Center, New York, New York
  - Montefiore-Einstein Center for Cancer Care, New York, New York
  - University of Virginia Health system, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No